CLINICAL TRIAL: NCT00095914
Title: Randomized, Crossover, Pharmacokinetic Study Of Paclitaxel (Taxol) And ABI-007 (A Cremophor EL-Free, Protein Stabilized, Nanoparticle Paclitaxel) In Patients With Advanced Solid Tumors
Brief Title: Paclitaxel and ABI-007 in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 040280; 04-C-0280; ABI-CA019; CDR0000393782; NCT00092261 (obsolete NCT alias)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Paclitaxel; Taxes

INTERVENTIONS:
Drug: paclitaxel
Drug: paclitaxel albumin-stabilized nanoparticle formulation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and ABI-007, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining paclitaxel with ABI-007 may kill more tumor cells.

PURPOSE: Randomized phase I trial to study the effectiveness of combining paclitaxel with ABI-007 in treating patients who have locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether a change in the formulation alters the pharmacokinetic profile of paclitaxel in the plasma of patients with incurable locally advanced or metastatic solid tumors treated with ABI-007 and paclitaxel.

Secondary

* Correlate pharmacokinetic data of this regimen with decrease in the neutrophil count at nadir in these patients.
* Determine the intra- and interindividual pharmacokinetic variability of ABI-007 in these patients.
* Determine protein binding of paclitaxel via measurement of α-1-acid glycoprotein and serum albumin levels in patients treated with this regimen.

OUTLINE: This is a randomized, pilot study.

* Courses 1 and 2: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive paclitaxel IV over 3 hours on day 1 and ABI-007 IV over 30 minutes on day 22.
  * Arm II: Patients receive ABI-007 IV over 30 minutes on day 1 and paclitaxel IV over 3 hours on day 22.
* Courses 3 and beyond: All patients receive ABI-007 IV over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant solid tumor

  * Considered incurable
  * Locally advanced or metastatic disease
* Likely to be responsive to taxane-based therapy

  * Patients who are refractory to prior paclitaxel are ineligible
* No symptomatic or untreated brain metastasis or carcinomatous meningitis

  * No patients who are unable to remain free of corticosteroid therapy for > 4 weeks due to CNS disease
* No previously untreated locally advanced breast cancer
* No hematologic malignancy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* ALT and AST ≤ 1.5 times upper limit of normal

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* LVEF ≥ 40%
* No clinical signs or symptoms of heart failure
* No symptomatic congestive heart failure
* No unstable angina pectoris

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study participation
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to paclitaxel (e.g., docetaxel, Cremophor^® EL [CrEL], polysorbate 80 [Tween 80], or CrEL-containing medications [e.g., cyclosporine])
* No history of seizure disorder requiring anticonvulsant therapy
* No active serious infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy
* No concurrent filgrastim (G-CSF) during courses 1 and 2

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 2 weeks since prior hormonal therapy
* Concurrent luteinizing hormone-releasing hormone agonists for prostate cancer allowed

Radiotherapy

* At least 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* More than 2 weeks since prior drugs, herbal preparations, or dietary supplements known to influence CYP3A4 (e.g., phenytoin, rifampin, Hypericum perforatum [St. John's wort], garlic supplements, or grapefruit juice) and/or CYP2C8
* No concurrent substances known or likely to interfere with the pharmacokinetics of paclitaxel (e.g., verapamil or cyclosporine)
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-09; Primary Completion 2007-05 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William D. Figg, PharmD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States